CLINICAL TRIAL: NCT05859438
Title: INcorporating VoIce AcTivated Communication Aids Into Everyday Communication
Acronym: INVITE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sheffield (Other)
Collaborators: Barnsley Hospital NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 171440
Record Dates: First submitted 2023-04-20; First posted 2023-05-16 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2024-12

CONDITIONS: Dysarthria
MeSH Terms: conditions — Dysarthria

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intervention group (Experimental)
  Interventions: Other: Communication aid support

INTERVENTIONS:
Other: Communication aid support — Support to use voice input voice output communication aids

SUMMARY:
Dysarthria is a speech disorder resulting in speech that is slow, slurred and difficult to understand, limiting a person's opportunities to study, work, and develop relationships.

People with dysarthria often use communication aids to help them to communicate creating spoken messages using a keyboard, touchscreen or joystick. Communication aids can increase independence but are often too slow to keep pace with normal conversation.

Developments in speech recognition technology have led to apps which can learn to recognise a set of words or sounds spoken by the individual with dysarthria, and connect these with a clear spoken output. The investigator's previous research provides some evidence that these voice input communication apps may be faster than traditional communication aids. This study aims to find out who can benefit from this technology, and what support they will need to use it successfully. This information can be used by professionals involved in providing communication aids, and will help the investigators to plan further research into their effectiveness.

This research has two phases:

1. 20-30 individuals with dysarthria will be asked to use a voice input communication app for 6 months. The investigator's will collect information on whether VocaTempo improves their communication, and helps participants to reach their goals.
2. Focus groups will be held with professionals involved in providing and supporting people with communication aids, to understand factors affecting their ability to provide the support identified as needed in part 1 of the research.

The investigators have a panel of communication aid users, who are advising and contributing throughout the study, for example, helping the investigators to identify informal support networks to recruit participants from. The investigators will let people know about the findings through support groups used by people with dysarthria, publications read by people involved in providing communication aids, and academic papers and conferences.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years of age
* Moderately or severely dysarthric (identified using the Frenchay Dysarthria assessment
* Minimum of 2 distinct vocalisations over which they have voluntary control
* Able to give informed consent and take part in interviews with appropriate communication support (scores level 1-3 on consent support tool)
* Communicates predominantly in English

Exclusion Criteria:

* They have significant cognitive impairment and are unable to give informed consent on their own behalf or actively take part in interviews (tested using the Consent Support Tool, scoring at level 4), or are unable to use a communication aid.
* They have no controlled vocalisations.
* They have dysarthria as a result of a progressive condition

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-05-31 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Goal Attainment Scale (measuring change between time points of distance from goal) | Baseline, 3 and 6 months
  Measures attainment of participant defined goals.

SECONDARY OUTCOMES:
Pragmatic Profile of Everyday Communication Skills in Adults (measuring change between time points of pragmatic communication) | Baseline, 3 and 6 months.
  Assesses pragmatic language use

OTHER OUTCOMES:
Speed of Communication by measuring time taken to speak out phrase with device - measuring change between timepoints. | 3 and 6 months
  Measuring speed of communicating with communication aid
System Usability Scale (measuring change between time points) | 3 and 6 months
  Questionnaire asking about usability of communication aid
Semi-structured interview | Baseline
  Conversation to ascertain participants experience
Semi-structured interview | 3 months
  Conversation to ascertain participants experience
Semi-structured interview | 6 months
  Conversation to ascertain participants experience
Participant diary (emails between participant and research which will be used as qualitative data). | 6 months
  Email diary

CONTACTS AND LOCATIONS:
Overall Officials: Kate Fryer, Principal Investigator — University of Sheffield
Locations (1):
- Barnsley Hospital NHS Foundation Trust, Barnsley, United Kingdom

IPD SHARING:
Plan to Share IPD: No